CLINICAL TRIAL: NCT07112989
Title: Development of Innovative Preclinical Ex Vivo Models for the Study of Sarcomas and Metastases From Solid Tumors
Acronym: PREMOD
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 477/2024/Sper/IOR
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Bone and Soft Tissue Tumors; Bone Metastases From Solid Tumors; Lung Metastases
Keywords: Sarcomas; Bone metastases; Lung metastases; Preclinical models
MeSH Terms: conditions — Soft Tissue Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue and peripheral blood samples will be collected from participants during standard diagnostic or therapeutic procedures. Tissue samples may include material from biopsies or surgical resections (primary tumors, recurrences, or metastases) that is in excess of what is needed for clinical diagnosis. Blood samples will be collected at predefined timepoints (e.g., diagnosis, post-treatment, follow-up) and processed to isolate serum, plasma, and mononuclear cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Sarcoma or Bone and Lung Metastases from Solid Tumors: This group includes male and female patients aged 0-85 years diagnosed with sarcomas or with bone or lung metastases from solid tumors and undergoing in surgical removal of the tumor or performing a biopsy. Only patients whose resection will provide sufficient tumor tissue that exceed what is necessary for pathological diagnosis characterization and banking will be enrolled.

SUMMARY:
The goal of this observational study is to learn how tumor tissue and blood samples from patients with sarcomas or metastases can be used to create laboratory models that help researchers study cancer behavior and test new treatments. Participants diagnosed with sarcoma or with bone or lung metastases from solid tumors will donate leftover tumor tissue and blood collected during their regular medical care. These samples will be used in the lab to build 3D models of the tumor, test drugs, and identify genetic and molecular markers. No treatments or procedures will be given as part of the study.

DETAILED DESCRIPTION:
PREMOD is a prospective, observational, preclinical study designed to develop and optimize innovative tumor models derived from patients diagnosed with sarcomas or with bone/lung metastases from solid tumors. These models include tumor explants, primary cultures, spheroids, scaffold-based 3D cultures, 3D bioprinted models, alginate capsules, and the chorioallantoic membrane (CAM) model.

Study Objectives

Primary Objective:

- To develop and optimize innovative preclinical models for study sarcomas and metastases.

Secondary Objectives:

* Identification of markers that can be proposed as possible therapeutic targets for rational use of drugs;
* Identification of circulating biomarkers capable of monitoring (and predicting) disease progression;
* Identification of circulating biomarkers predictive of toxicity to treatments;
* Identification of innovative therapeutic strategies for the treatment of sarcomas and metastases; Study Tasks and Scope

The study includes four main research tasks:

Task 1: Optimization of innovative ex vivo preclinical models. Develop different preclinical tumour models from patient-derived tissue. Each model is optimised to study specific features of tumour biology and its interactions with the microenvironment. Success in developing the models is assessed using defined criteria such as cell viability and model reproducibility.

Task 2: Study of the natural history of sarcomas and metastases. The developed models are used to investigate tumour cell behaviour, including growth, invasiveness and interaction with the microenvironment and molecular profiling.

Task 3: Drug screening. Patient-derived models are used to evaluate the efficacy of conventional or innovative drugs as single agents or in combination. Locoregional treatments (e.g., electrochemotherapy, cryotherapy, thermoablation) may also be tested.

Task 4: Identification of prognostic markers, or predictors of response or toxicity to treatment.

Biological samples are analyzed to identify prognostic and predictive biomarkers, including circulating markers and genetic polymorphisms linked to treatment response or toxicity.

Study Size and Duration Approximately 125 patients (including about 90 with sarcoma and 35 with bone or lung metastasis from solid tumor) will be enrolled over a 5-year recruitment period (25 per year), with a total study duration of 7 years. No investigational treatments are administered to participants. All experimental work is conducted ex vivo using donated biological material.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) diagnosed with sarcoma or with bone or lung metastases from solid tumors
* Age between 0 and 85 years
* Availability of sufficient and adequate biological material (tumor tissue and/or blood)
* Signed informed consent for biobanking (BIOTUM)
* Signed informed consent for use of tissue and blood samples in this study

Exclusion Criteria:

* Diagnosis other than sarcoma or metastases from solid tumors
* Missing signed informed consent(s)

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes male and female patients aged 0 to 85 years who have been diagnosed with sarcoma or with bone or lung metastases from solid tumors. Only patients whose resection will provide sufficient tumor tissue that exceed what is necessary for pathological diagnosis characterization and banking will be enrolled. Participation is voluntary and requires signed informed consent for biobanking and for the use of biological samples. Approximately 125 patients are expected to be enrolled over five years (around 90 with sarcoma and 35 with metastatic disease).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2031-09-23 (Estimated); Study Completion 2031-09-23 (Estimated)

PRIMARY OUTCOMES:
Number of tumor samples enabling the development of at least three preclinical models | 7 years
  Number of patient-derived tumor samples that allow the successful development of at least three distinct preclinical models (e.g., spheroids, explants, scaffold-based cultures, or bioprinted constructs). This outcome assesses the feasibility and robustness of the tissue-based modeling approach.

SECONDARY OUTCOMES:
Evaluation of the quality of the models | 7 years
  Assessment of cell viability in the developed preclinical models. A model will be considered successful if at least 80% of cells are viable after 7 days of in vitro culture, as measured by standard viability assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy